CLINICAL TRIAL: NCT02182336
Title: Evaluation of the Effects of Single Oral Dose and Multiple Oral Doses of BI 201335 NA on Cytochrome P450 and P-glycoprotein Activity Using a Probe Drug Cocktail. An Open-label, Single-arm Phase I Study in Healthy Human Volunteers
Brief Title: Effects of BI 201335 NA on Cytochrome P450 and P-glycoprotein Activity Using a Probe Drug Cocktail in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1220.32
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Caffeine; Warfarin; Vitamin K; Omeprazole; Dextromethorphan; Digoxin

ARMS (1):
- BI 201335 NA (Experimental)
  Interventions: Drug: BI 201335 NA; Drug: Caffeine; Drug: Warfarin sodium; Drug: Vitamin K; Drug: Omeprazole; Drug: Dextromethorphan hydrobromide; Drug: Midazolam HCl solution; Drug: Midazolam HCl oral syrup; Drug: Digoxin

INTERVENTIONS:
Drug: BI 201335 NA — 1. 480 mg BI 201335 NA in the morning, 240 mg BI 201335 NA in the evening of day 10
  2. 240 mg BI 201335 NA bid from day 11 to 23
Drug: Caffeine — days 1, 10 and 19
Drug: Warfarin sodium — days 1, 10 and 19
Drug: Vitamin K — days 1, 10 and 19
Drug: Omeprazole — days 1, 10 and 19
Drug: Dextromethorphan hydrobromide — days 1, 10 and 19
Drug: Midazolam HCl solution — Days 3 and 21
Drug: Midazolam HCl oral syrup — days 1, 10 and 19
Drug: Digoxin — Days 2 and 20

SUMMARY:
The objective of this trial was to quantify the effect of oral single-dose (480 mg) and steady-state BI 201335 NA (240 mg BID) on intestinal and hepatic cytochrome P450 (CYP) and P-glycoprotein (P-gp) probe drugs as a means of predicting drug interactions. The AUCs for the probe drugs caffeine, warfarin, omeprazole, dextromethorphan, midazolam, and digoxin were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation
* Healthy males and female subjects age ≥18 to ≤55 years and according to the following criteria:

  * Complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead EKG (electrocardiogram)(including determination of QTcB, and QtcF intervals), and clinical laboratory tests; all with acceptable findings
* Weighing at least 50 kg, and BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Volunteers must not leave the research unit, during the days of over-night stays, which include the periods from evening of Day-1 to morning of Day 5, and evening of Day 9 to morning of Day 24
* Volunteers must be willing to complete all study-related activities

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and EKG) deviating from normal and of clinical relevance, as assessed by the investigator
* Active diseases of the gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, musculoskeletal, immunologic, rheumatologic, hormonal, neurological system, cancer, or bleeding disorders that require current medical treatment, may be unstable, or may be exacerbated by participation in the study
* Any evidence of a clinically relevant concomitant disease, which is not defined in the exclusion criteria 2 above, including but not limited to relevant chronic or acute infection
* Surgery of the gastrointestinal tract (except appendectomy and endoscopic removal of colon polyps)
* History or presence of allergy to any of the study drugs (e.g., BI 201335 NA, caffeine, warfarin, vitamin K, omeprazole, dextromethorphan, digoxin, midazolam, omeprazole) or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* Concomitant drugs, nutraceuticals, and herbal remedies that in the opinion of the investigator (in consultation with the BI medical monitor or pharmacokineticist), would interfere with either the absorption, distribution or metabolism of BI 201335 NA, or other study drugs
* Use of drugs, which might reasonably influence the results of the trial or that prolong the QT/QTc interval within 30 days prior to screening until trial completion
* Use of any investigational drug within 30 days prior to enrollment; or the planned usage of any investigational drug during the course of the current study
* Smoking (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to abstain from alcohol from day of screening to 7 days after last study drug administration.
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial
* Any laboratory value outside the reference range that is of clinical relevance at screening, according to the judgment of the investigator, and in consultation with the clinical monitor
* Known elevated liver enzymes in past with any compound (experimental or marketed)
* Concomitant administration of any food product known to alter P450 enzyme or P-gp activity such as grapefruit juice, Seville oranges, St. John's Wort
* Concomitant administration of any drug that could affect bleeding (e.g., aspirin, clopidogrel, ticlopidine, warfarin in addition to the studied warfarin dose, heparin, low-molecular weight heparin)
* Concomitant administration of oral contraceptives (may be included with 7-day washout period)
* Inadequate venous access
* Renal or hepatic insufficiency
* A marked baseline prolongation of QT/QTc interval e.g., repeated demonstration of a QTcF, or QTcB interval >450 ms)
* Infection with hepatitis B (HBV), or hepatitis C virus (HCV), defined as either being hepatitis B surface antigen and /or hepatitis B core antibody positive, or hepatitis C antibody positive)
* Positive Enzyme-linked immunosorbent assay (ELISA) for Human Immunodeficiency Virus (HIV)-1 or HIV-2
* Fasting screening laboratory testing with direct bilirubin within the normal range and elevated total bilirubin, defined as 30% above the upper limit of normal
* For female subjects:

  * Pregnancy or planning to become pregnant within 2 months of study completion
  * Positive pregnancy test at screening visit
  * No adequate contraception, e.g., sterilisation, IUD (intrauterine device), have not been using a barrier method of contraception for at least 3 months prior to participation in the study
  * Are not willing or are unable to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and up to 2 months after completion/termination of the trial
  * Lactation period with active breastfeeding from time of screening to 30 days after end of trial visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) 0-24h of caffeine | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 hours after treatment on days 1, 10 and 19
AUC0-120h of Warfarin | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours after treatment on days 1, 10 and 19
AUC0-24h of Omeprazole | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 hours after treatment on days 1, 10 and 19
AUC0-24h of Dextromethorphan | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 hours after treatment on days 1, 10 and 19
AUC0-24h of Midazolam IV | Pre-dose and 0.08, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours after treatment on days 3 and 21
AUC0-24h of Midazolam oral | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 hours after treatment on days 1, 10 and 19
AUC0-96h of Digoxin | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours after treatment on days 2 and 20

SECONDARY OUTCOMES:
AUC of caffeine | Baseline and day 1, day 1 and day 19
Cmax (Maximum Plasma Concentration after a single dose) of caffeine | Baseline and day 1, baseline and day 19
Ct (Plasma concentration at a given time t after a single dose) of caffeine | Baseline and day 1, baseline and day 19
tmax (Time of Maximum Concentration after a single dose) of caffeine | Baseline and day 1, baseline and day 19
CL/F (Oral Clearance after a single dose) of caffeine | Baseline and day1, baseline and day 19
t1/2 (Apparent Terminal Half-Life) of caffeine | Baseline and day 1, baseline and day 19
AUC of Warfarin | Baseline and day 1, day 1 and day 19
Cmax of Warfarin | Baseline and day 1, day 1 and day 19
Ct of Warfarin | Baseline and day 1, day 1 and day 19
tmax of Warfarin | Baseline and day 1, day 1 and day 19
CL/F of Warfarin | Baseline and day 1, day 1 and day 19
t1/2 of Warfarin | Baseline and day 1, day 1 and day 19
AUC of Omeprazole | Baseline and day 1, day 1 and day 19
Cmax of Omeprazole | Baseline and day 1, day 1 and day 19
Ct of Omeprazole | Baseline and day 1, day 1 and day 19
tmax of Omeprazole | Baseline and day 1, day 1 and day 19
CL/F of Omeprazole | Baseline and day 1, day 1 and day 19
t1/2 of Omeprazole | Baseline and day 1, day 1 and day 19
AUC of Dextromethorphan | Baseline and day 1, day 1 and day 19
Cmax of Dextromethorphan | Baseline and day 1, day 1 and day 19
Ct of Dextromethorphan | Baseline and day 1, day 1 and day 19
tmax of Dextromethorphan | Baseline and day 1, day 1 and day 19
CL/F of Dextromethorphan | Baseline and day 1, day 1 and day 19
t1/2 of Dextromethorphan | Baseline and day 1, day 1 and day 19
AUC of Midazolam IV | Baseline and day 1, day 1 and day 19
Cmax of Midazolam IV | Baseline and day 1, day 1 and day 19
Ct of Midazolam IV | Baseline and day 1, day 1 and day 19
tmax of Midazolam IV | Baseline and day 1, day 1 and day 19
CL/F of Midazolam IV | Baseline and day 1, day 1 and day 19
t1/2 of Midazolam IV | Baseline and day 1, day 1 and day 19
AUC of Midazolam oral | Baseline and day 1, baseline and day 19
Cmax of Midazolam oral | Baseline and day 1, baseline and day 19
Ct of Midazolam oral | Baseline and day 1, baseline and day 19
tmax of Midazolam oral | Baseline and day 1, baseline and day 19
CL/F of Midazolam oral | Baseline and day 1, baseline and day 19
t1/2 of Midazolam oral | Baseline and day 1, baseline and day 19
AUC of Digoxin | Baseline and day 1, baseline and day 19
Cmax of Digoxin | Baseline and day 1, baseline and day 19
Ct of Digoxin | Baseline and day 1, baseline and day 19
tmax of Digoxin | Baseline and day 1, baseline and day 19
CL/F of Digoxin | Baseline and day 1, baseline and day 19
t1/2 of Digoxin | Baseline and day 1, baseline and day 19
AUCτ,N (Uniform Dosing Interval τ Following the Nth Dose) of BI201335 NA | Day 10
AUCτ,ss,N of BI201335 NA | Day 19
Cmax,N of BI 201335 NA | Day 10
Cmax,ss,N of BI 201335 NA | Day 19
tmax,N of BI 201335 NA | Day 10
tmax,ss,N of BI 201335 NA | Day 19
Cmin,N of BI 201335 NA | Day 10
Cmin,ss,N of BI 201335 NA | Day 19
CL/F,ss,N of BI 201335 NA | Day 19
Urinary metabolic ratios of the analyte of first-day and steady state | up to day 19